CLINICAL TRIAL: NCT01981187
Title: Modular Phase II Study to Link Targeted Therapy to Patients With Pathway Activated Tumors: Module 4 - LGX818 for Patients With BRAFV600 Mutated Tumors
Brief Title: LGX818 for Patients With BRAFV600 Mutated Tumors
Acronym: SIGNATURE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow enrollment and lack of response observed during the enrollment period, the Sponsor decided to close study enrollment early on 28 January 2015
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: CLGX818AUS03; C4221021 (Other: Alias Study Number)
Record Dates: First submitted 2013-11-05; First posted 2013-11-11 (Estimated); Results first posted 2021-03-26 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Solid Tumor; Hematologic Malignancies
MeSH Terms: conditions — Hematologic Neoplasms | interventions — encorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LGX818 (Experimental): LGX818 will be dosed on a flat scale of 300 mg (e.g., 3 x 100 mg capsules) once daily on a continuous dosing cycle. A complete treatment cycle is defined as 28 days. There will be no breaks between dosing cycles.
  Interventions: Drug: LGX818

INTERVENTIONS:
Drug: LGX818 — LGX818 will be dosed on a flat scale of 300 mg (e.g., 3 x 100 mg capsules) once daily on a continuous dosing cycle. A complete treatment cycle is defined as 28 days. There will be no breaks between dosing cycles.

SUMMARY:
The purpose of this signal seeking study is to determine whether treatment with LGX818 demonstrates sufficient efficacy in select pathway-activated solid tumors and/or hematologic malignancies to warrant further study

ELIGIBILITY:
Inclusion Criteria

* Patient has a confirmed diagnosis of a select solid tumor (except with a primary diagnosis of melanoma and colorectal cancer (CRC)) or hematologic malignancies and is in need of treatment because of progression or relapse.
* Patient's tumor has been evaluated and pre-identified as having a tumor with a BRAFV600 mutation at a CLIA certified laboratory.
* Patient must have received at least one prior treatment for recurrent, metastatic and /or locally advanced disease and for whom no standard therapy options are anticipated to result in a durable remission.
* Patient must have progressive and measurable disease per RECIST 1.1. or other appropriate hematological response criteria.
* Patient has an Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1

Exclusion Criteria:

* Patient has received prior treatment with LGX818.
* Patients with Central Nerve System (CNS) metastasis or leptomeningeal carcinomatosis.
* Patient has received chemotherapy or other anticancer therapy ≤ 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug.
* Patients with acute or chronic pancreatitis.
* Patients with impaired cardiac function or clinically significant cardiac diseases.
* Patients with another primary malignancy within 3 years prior to starting study treatment, with the exception of adequately treated basal cell carcinoma, squamous cell carcinoma or other non-melanomatous skin cancer, or in-situ carcinoma of the uterine cervix.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01-14 (Actual); Primary Completion 2015-09-01 (Actual); Study Completion 2015-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (13):
- United States (13):
  - Alabama Oncology St. Vincent's Birmingham, Birmingham, Alabama
  - Highlands Oncology Group Highlands Oncology Group (22), Fayetteville, Arkansas
  - Yale University School of Medicine Smilow Cancer Hospital, New Haven, Connecticut
  - Whittingham Cancer Center Norwalk Hospital, Norwalk, Connecticut
  - Florida Cancer Specialists Florida Cancer Specialists (31, Fort Myers, Florida
  - Lurie Children's Hospital of Chicago Developmental Therapeutics, Chicago, Illinois
  - Comprehensive Cancer Centers of Nevada CCC of Nevada (1), Las Vegas, Nevada
  - Genesis Cancer Services, Zanesville, Ohio
  - University of Pennsylvania Presbyterian Medical Center University of Pennsylvania, Philadelphia, Pennsylvania
  - Sanford Research Sanford Health, Sioux Falls, South Dakota
  - Oncology Consultants Oncology Group, Houston, Texas
  - Utah Cancer Specialists Utah Cancer Specialists (11), Salt Lake City, Utah
  - Shenandoah Oncology Shenadoah Oncology (2), Winchester, Virginia

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

RESULTS

PARTICIPANT FLOW:
Groups:
- LGX818 (Encorafenib): Participants received an oral dose of 300 mg of LGX818 (Encorafenib) capsules (3 capsules of 100 mg) once daily in each cycle (1 cycle = 28 days) until disease progression, unacceptable toxicity, death or discontinuation from study treatment for any other reason. Maximum study treatment exposure was approximately of 12 months and participants were followed up to 13.3 months approximately.
Period: Overall Study
Arm/Group | LGX818 (Encorafenib)
Started | 12
Completed | 0
Not Completed | 12
Not completed — Participant/guardian decision | 2
Not completed — Physician Decision | 1
Not completed — Disease progression | 2
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who received at least one dose of study drug.
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.6 (11.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) for Solid Tumors as Per Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Description: CBR for solid tumors was defined as percentage of participants with complete response (CR) or partial response (PR), or stable disease (SD) for greater than or equal to (>=) 16 weeks. As per RECIST v1.1, CR was defined as disappearance of all target and non-target lesions and normalization of tumor markers. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease, taking as reference the smallest sum diameters while on study. PD was defined as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline.
Time Frame: Up to 13.3 months
Population: The full analysis set included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
percentage of participants | 25 [5.5 to 57.2]

2. Secondary Outcome: Overall Response Rate (ORR) for Solid Tumors as Per RECIST Version 1.1
Description: ORR for solid tumors was defined as the percentage of participants achieving an overall best response of CR or PR as assessed per RECIST version 1.1. CR was defined as disappearance of all target and non-target lesions and normalization of tumor markers. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as least a 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the first dose study treatment until the first documented CR or PR (maximum up to 13.3 months)
Population: The full analysis set included all participants who received at least one dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
percentage of participants | 0 [0.0 to 26.5]

3. Secondary Outcome: Progression-Free Survival (PFS) for Solid Tumors as Per RECIST Version 1.1
Description: PFS for solid tumors was defined as the time from the date of first dose of study drug to the date of first documented disease progression (PD) or relapse or death due to any cause within 30 days of the last dose. PD was defined as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. Participants who had no event were censored at the date of last adequate tumor assessment.
Time Frame: From the date of first dose until the first documentation of PD, relapse, censored date or death, whichever occurred first (maximum up to 13.3 months)
Population: The full analysis set included all participants who received at least one dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
months | NA [1.8 to NA] — Median and upper limit of 95% CI were not estimable due to low number of participants with an event.

4. Secondary Outcome: Overall Survival (OS) for Solid Tumors
Description: OS for solid tumors was defined as the time from the date of first dose of study drug to the date of death due to any cause. For participants who were alive at the time of analysis, the data was censored at the date of last contact.
Time Frame: From date of the first dose until the date of death, censored date (maximum up to 13.3 months)
Population: The full analysis set included all participants who received at least one dose of study drug.
Measure: Median (Full Range); unit: months
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
months | 13.3 [8.4 to 13.3]

5. Secondary Outcome: Duration of Response (DOR) for Solid Tumors as Per RECIST Version 1.1
Description: DOR for solid tumors was defined as the time from the first documented response (CR or PR) to the date of first documented PD or relapse or death due to any cause, whichever occurred first. As per RECIST v1.1, CR was defined as disappearance of all target and non-target lesions and normalization of tumor markers. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. PR was defined as least a 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as at least a 20% increase in the sum of diameter of all measured target lesions, taking as reference the smallest sum of diameter of all target lesions recorded at or after baseline. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: From first documentation of response to first documentation of PD or relapse or death (maximum up to 13.3 months)
Population: Data for this outcome measure was not analyzed due to low overall response rate among participants.
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 0

6. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) Graded According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03
Description: Adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. As per NCI-CTCAE version 4.03, severity was graded as Grade 1: asymptomatic/mild symptoms, clinical/diagnostic observations only, intervention not indicated; Grade 2: moderate, minimal, local/noninvasive intervention indicated, limiting age-appropriate instrumental activities of daily life (ADL); Grade 3: severe/medically significant but not immediately life-threatening, hospitalization/prolongation of existing hospitalization indicated, disabling, limiting self-care ADL; Grade 4: life-threatening consequence, urgent intervention indicated. TEAE was defined as event with onset dates occurring during the on-treatment period. CTCAE Grade 5 (death) was not used in this study.
Time Frame: Screening up to 30 days after the last dose of study treatment (maximum up to 13.3 months)
Population: The safety set included all participants who received at least one dose of study treatment and had at least one post-baseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
Participants
  Grade 1 | 0
  Grade 2 | 2
  Grade 3 | 10
  Grade 4 | 0

7. Secondary Outcome: Change From Baseline in Systolic and Diastolic Blood Pressure
Description: Change from baseline in systolic and diastolic blood pressure in millimeter of mercury (mmHg) in sitting position was reported.
Time Frame: Baseline, Day 1 of Cycle 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 (each cycle of 28 days), and End of treatment (up to 7 days after study treatment discontinuation)
Population: The safety set included all participants who received at least one dose of study treatment and had at least one post-baseline safety assessment. Here 'number analyzed' signifies number of participants evaluable for each specified row.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
mmHg
  Systolic Blood Pressure: Baseline | 129.4 (17.33)
  Systolic Blood Pressure: Change at Cycle 2, Day 1: number analyzed (Participants) | 8
  Systolic Blood Pressure: Change at Cycle 2, Day 1 | 2.4 (4.34)
  Systolic Blood Pressure: Change at Cycle 3, Day 1: number analyzed (Participants) | 5
  Systolic Blood Pressure: Change at Cycle 3, Day 1 | 4.0 (23.56)
  Systolic Blood Pressure: Change at Cycle 4, Day 1: number analyzed (Participants) | 4
  Systolic Blood Pressure: Change at Cycle 4, Day 1 | -0.3 (14.52)
  Systolic Blood Pressure: Change at Cycle 5, Day 1: number analyzed (Participants) | 4
  Systolic Blood Pressure: Change at Cycle 5, Day 1 | 7.8 (11.32)
  Systolic Blood Pressure: Change at Cycle 6, Day 1: number analyzed (Participants) | 3
  Systolic Blood Pressure: Change at Cycle 6, Day 1 | -5.3 (18.01)
  Systolic Blood Pressure: Change at Cycle 7, Day 1: number analyzed (Participants) | 3
  Systolic Blood Pressure: Change at Cycle 7, Day 1 | 0.0 (12.49)
  Systolic Blood Pressure: Change at Cycle 8, Day 1: number analyzed (Participants) | 2
  Systolic Blood Pressure: Change at Cycle 8, Day 1 | 1.5 (4.95)
  Systolic Blood Pressure: Change at Cycle 9, Day 1: number analyzed (Participants) | 1
  Systolic Blood Pressure: Change at Cycle 9, Day 1 | 2.0 (NA) — Standard deviation was not estimated due to single participant.
  Systolic Blood Pressure: Change at Cycle 10, Day 1: number analyzed (Participants) | 1
  Systolic Blood Pressure: Change at Cycle 10, Day 1 | 9.0 (NA) — Standard deviation was not estimated due to single participant.
  Systolic Blood Pressure: Change at Cycle 11, Day 1: number analyzed (Participants) | 1
  Systolic Blood Pressure: Change at Cycle 11, Day 1 | 10.0 (NA) — Standard deviation was not estimated due to single participant.
  Systolic Blood Pressure: Change at Cycle 12, Day 1: number analyzed (Participants) | 1
  Systolic Blood Pressure: Change at Cycle 12, Day 1 | 15.0 (NA) — Standard deviation was not estimated due to single participant.
  Systolic Blood Pressure: Change at End of Treatment: number analyzed (Participants) | 9
  Systolic Blood Pressure: Change at End of Treatment | 8.7 (18.95)
  Diastolic Blood Pressure: Baseline | 78.1 (9.33)
  Diastolic Blood Pressure: Change at Cycle 2, Day 1: number analyzed (Participants) | 8
  Diastolic Blood Pressure: Change at Cycle 2, Day 1 | -0.1 (8.46)
  Diastolic Blood Pressure: Change at Cycle 3, Day 1: number analyzed (Participants) | 5
  Diastolic Blood Pressure: Change at Cycle 3, Day 1 | 1.4 (11.26)
  Diastolic Blood Pressure: Change at Cycle 4, Day 1: number analyzed (Participants) | 4
  Diastolic Blood Pressure: Change at Cycle 4, Day 1 | -1.3 (5.62)
  Diastolic Blood Pressure: Change at Cycle 5, Day 1: number analyzed (Participants) | 4
  Diastolic Blood Pressure: Change at Cycle 5, Day 1 | -0.5 (4.12)
  Diastolic Blood Pressure: Change at Cycle 6, Day 1: number analyzed (Participants) | 3
  Diastolic Blood Pressure: Change at Cycle 6, Day 1 | -0.7 (8.33)
  Diastolic Blood Pressure: Change at Cycle 7, Day 1: number analyzed (Participants) | 3
  Diastolic Blood Pressure: Change at Cycle 7, Day 1 | 1.7 (9.71)
  Diastolic Blood Pressure: Change at Cycle 8, Day 1: number analyzed (Participants) | 2
  Diastolic Blood Pressure: Change at Cycle 8, Day 1 | 1.0 (4.24)
  Diastolic Blood Pressure: Change at Cycle 9, Day 1: number analyzed (Participants) | 1
  Diastolic Blood Pressure: Change at Cycle 9, Day 1 | 0.0 (NA) — Standard deviation was not estimated due to single participant.
  Diastolic Blood Pressure: Change at Cycle 10, Day 1: number analyzed (Participants) | 1
  Diastolic Blood Pressure: Change at Cycle 10, Day 1 | 9.0 (NA) — Standard deviation was not estimated due to single participant.
  Diastolic Blood Pressure: Change at Cycle 11, Day 1: number analyzed (Participants) | 1
  Diastolic Blood Pressure: Change at Cycle 11, Day 1 | 5.0 (NA) — Standard deviation was not estimated due to single participant.
  Diastolic Blood Pressure: Change at Cycle 12, Day 1: number analyzed (Participants) | 1
  Diastolic Blood Pressure: Change at Cycle 12, Day 1 | 0.0 (NA) — Standard deviation was not estimated due to single participant.
  Diastolic Blood Pressure: Change at End of Treatment: number analyzed (Participants) | 9
  Diastolic Blood Pressure: Change at End of Treatment | 4.7 (12.12)

8. Secondary Outcome: Change From Baseline in Sitting Pulse Rate
Description: Change from baseline in pulse rate in beats per minute (bpm) in sitting position was reported.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
bpm
  Baseline | 84.8 (18.17)
  Change at Cycle 2, Day 1: number analyzed (Participants) | 8
  Change at Cycle 2, Day 1 | 4.9 (8.18)
  Change at Cycle 3, Day 1: number analyzed (Participants) | 5
  Change at Cycle 3, Day 1 | -1.2 (18.67)
  Change at Cycle 4, Day 1: number analyzed (Participants) | 4
  Change at Cycle 4, Day 1 | -19.0 (23.86)
  Change at Cycle 5, Day 1: number analyzed (Participants) | 4
  Change at Cycle 5, Day 1 | -5.0 (4.24)
  Change at Cycle 6, Day 1: number analyzed (Participants) | 3
  Change at Cycle 6, Day 1 | -10.3 (8.33)
  Change at Cycle 7, Day 1: number analyzed (Participants) | 3
  Change at Cycle 7, Day 1 | -4.3 (16.86)
  Change at Cycle 8, Day 1: number analyzed (Participants) | 2
  Change at Cycle 8, Day 1 | -1.0 (42.43)
  Change at Cycle 9, Day 1: number analyzed (Participants) | 1
  Change at Cycle 9, Day 1 | -24.0 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 10, Day 1: number analyzed (Participants) | 1
  Change at Cycle 10, Day 1 | -25.0 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 11, Day 1: number analyzed (Participants) | 1
  Change at Cycle 11, Day 1 | -19.0 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 12, Day 1: number analyzed (Participants) | 1
  Change at Cycle 12, Day 1 | -23.0 (NA) — Standard deviation was not estimated due to single participant.
  Change at End of Treatment: number analyzed (Participants) | 9
  Change at End of Treatment | -2.7 (9.33)

9. Secondary Outcome: Change From Baseline in Body Temperature
Description: Change from baseline in body temperature in degree Celsius was reported.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: degree Celsius
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
degree Celsius
  Baseline | 36.7 (0.30)
  Change at Cycle 2, Day 1: number analyzed (Participants) | 8
  Change at Cycle 2, Day 1 | -0.1 (0.32)
  Change at Cycle 3, Day 1: number analyzed (Participants) | 5
  Change at Cycle 3, Day 1 | 0.0 (0.25)
  Change at Cycle 4, Day 1: number analyzed (Participants) | 4
  Change at Cycle 4, Day 1 | -0.3 (0.13)
  Change at Cycle 5, Day 1: number analyzed (Participants) | 4
  Change at Cycle 5, Day 1 | 0.0 (0.13)
  Change at Cycle 6, Day 1: number analyzed (Participants) | 3
  Change at Cycle 6, Day 1 | -0.4 (0.36)
  Change at Cycle 7, Day 1: number analyzed (Participants) | 3
  Change at Cycle 7, Day 1 | -0.4 (0.42)
  Change at Cycle 8, Day 1: number analyzed (Participants) | 2
  Change at Cycle 8, Day 1 | -0.4 (0.42)
  Change at Cycle 9, Day 1: number analyzed (Participants) | 1
  Change at Cycle 9, Day 1 | -0.5 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 10, Day 1: number analyzed (Participants) | 1
  Change at Cycle 10, Day 1 | -0.5 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 11, Day 1: number analyzed (Participants) | 1
  Change at Cycle 11, Day 1 | -0.8 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 12, Day 1: number analyzed (Participants) | 1
  Change at Cycle 12, Day 1 | -0.4 (NA) — Standard deviation was not estimated due to single participant.
  Change at End of Treatment: number analyzed (Participants) | 9
  Change at End of Treatment | -0.1 (0.38)

10. Secondary Outcome: Change From Baseline in Respiratory Rate
Description: Change from baseline in respiratory rate in breaths per minute was reported.
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
breaths per minute
  Baseline | 17.6 (1.31)
  Change at Cycle 2, Day 1: number analyzed (Participants) | 8
  Change at Cycle 2, Day 1 | 0.0 (1.41)
  Change at Cycle 3, Day 1: number analyzed (Participants) | 5
  Change at Cycle 3, Day 1 | 2.0 (4.47)
  Change at Cycle 4, Day 1: number analyzed (Participants) | 4
  Change at Cycle 4, Day 1 | -1.0 (1.15)
  Change at Cycle 5, Day 1: number analyzed (Participants) | 4
  Change at Cycle 5, Day 1 | -0.5 (1.00)
  Change at Cycle 6, Day 1: number analyzed (Participants) | 3
  Change at Cycle 6, Day 1 | 0.0 (2.00)
  Change at Cycle 7, Day 1: number analyzed (Participants) | 3
  Change at Cycle 7, Day 1 | 0.7 (1.15)
  Change at Cycle 8, Day 1: number analyzed (Participants) | 2
  Change at Cycle 8, Day 1 | -1.0 (1.41)
  Change at Cycle 9, Day 1: number analyzed (Participants) | 1
  Change at Cycle 9, Day 1 | 0.0 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 10, Day 1: number analyzed (Participants) | 1
  Change at Cycle 10, Day 1 | 0.0 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 11, Day 1: number analyzed (Participants) | 1
  Change at Cycle 11, Day 1 | 0.0 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 12, Day 1: number analyzed (Participants) | 1
  Change at Cycle 12, Day 1 | 1.0 (NA) — Standard deviation was not estimated due to single participant.
  Change at End of Treatment: number analyzed (Participants) | 9
  Change at End of Treatment | -0.1 (1.76)

11. Secondary Outcome: Change From Baseline in Body Weight
Description: Change from baseline in body weight in kilogram (Kg) was reported
Time Frame: as for outcome 7
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
Kg
  Baseline | 87.0 (21.77)
  Change at Cycle 2, Day 1: number analyzed (Participants) | 8
  Change at Cycle 2, Day 1 | -3.4 (2.48)
  Change at Cycle 3, Day 1: number analyzed (Participants) | 5
  Change at Cycle 3, Day 1 | -3.4 (2.77)
  Change at Cycle 4, Day 1: number analyzed (Participants) | 4
  Change at Cycle 4, Day 1 | -6.5 (3.85)
  Change at Cycle 5, Day 1: number analyzed (Participants) | 4
  Change at Cycle 5, Day 1 | -5.8 (3.96)
  Change at Cycle 6, Day 1: number analyzed (Participants) | 3
  Change at Cycle 6, Day 1 | -6.0 (4.57)
  Change at Cycle 7, Day 1: number analyzed (Participants) | 3
  Change at Cycle 7, Day 1 | -6.8 (5.96)
  Change at Cycle 8, Day 1: number analyzed (Participants) | 2
  Change at Cycle 8, Day 1 | -6.4 (4.81)
  Change at Cycle 9, Day 1: number analyzed (Participants) | 1
  Change at Cycle 9, Day 1 | -12.5 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 10, Day 1: number analyzed (Participants) | 1
  Change at Cycle 10, Day 1 | -10.3 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 11, Day 1: number analyzed (Participants) | 1
  Change at Cycle 11, Day 1 | -9.4 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 12, Day 1: number analyzed (Participants) | 1
  Change at Cycle 12, Day 1 | -9.0 (NA) — Standard deviation was not estimated due to single participant.
  Change at End of Treatment: number analyzed (Participants) | 9
  Change at End of Treatment | -3.7 (3.43)

12. Secondary Outcome: Number of Participants With Shifts From Baseline in Hematology and Serum Chemistry Laboratory Abnormalities
Description: Number of participants with shifts from baseline in hematology and serum chemistry laboratory parameters, were graded and reported as low, normal and high as assessed by Common terminology criteria for adverse events (CTCAE) v4.03. 'Low' refers to participants with values that were below lower limit of normal with no observation above the upper limit of normal; 'High' refers to participants with values that were above the upper limit of normal with no observation below the lower limit of normal; 'Low and High' refers to participants with values that were below the lower limit of normal and values that were above the upper limit of normal.
Time Frame: Baseline up to maximum of 30 days after the last dose of study treatment (up to 13.3 months)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
Participants
  Red Blood Cell Count, Low: number analyzed (Participants) | 11
  Red Blood Cell Count, Low | 5
  Red Blood Cell Count, Normal: number analyzed (Participants) | 11
  Red Blood Cell Count, Normal | 6
  Red Blood Cell Count, High: number analyzed (Participants) | 11
  Red Blood Cell Count, High | 0
  Hematocrit, Low: number analyzed (Participants) | 11
  Hematocrit, Low | 7
  Hematocrit, Normal: number analyzed (Participants) | 11
  Hematocrit, Normal | 4
  Hematocrit, High: number analyzed (Participants) | 11
  Hematocrit, High | 0
  Eosinophils, Low: number analyzed (Participants) | 10
  Eosinophils, Low | 0
  Eosinophils, Normal: number analyzed (Participants) | 10
  Eosinophils, Normal | 7
  Eosinophils, High: number analyzed (Participants) | 10
  Eosinophils, High | 3
  Basophils, Low: number analyzed (Participants) | 10
  Basophils, Low | 0
  Basophils, Normal: number analyzed (Participants) | 10
  Basophils, Normal | 9
  Basophils, High: number analyzed (Participants) | 10
  Basophils, High | 1
  Monocytes, Low: number analyzed (Participants) | 10
  Monocytes, Low | 0
  Monocytes, Normal: number analyzed (Participants) | 10
  Monocytes, Normal | 3
  Monocytes, High: number analyzed (Participants) | 10
  Monocytes, High | 7
  Neutrophils, Low: number analyzed (Participants) | 1
  Neutrophils, Low | 0
  Neutrophils, Normal: number analyzed (Participants) | 1
  Neutrophils, Normal | 0
  Neutrophils, High: number analyzed (Participants) | 1
  Neutrophils, High | 1
  Lymphocytes, Low: number analyzed (Participants) | 1
  Lymphocytes, Low | 0
  Lymphocytes, Normal: number analyzed (Participants) | 1
  Lymphocytes, Normal | 1
  Lymphocytes, High: number analyzed (Participants) | 1
  Lymphocytes, High | 0
  Blood Urea Nitrogen, Low: number analyzed (Participants) | 11
  Blood Urea Nitrogen, Low | 1
  Blood Urea Nitrogen, Normal: number analyzed (Participants) | 11
  Blood Urea Nitrogen, Normal | 8
  Blood Urea Nitrogen, High: number analyzed (Participants) | 11
  Blood Urea Nitrogen, High | 2
  Bicarbonate, Low: number analyzed (Participants) | 11
  Bicarbonate, Low | 2
  Bicarbonate, Normal: number analyzed (Participants) | 11
  Bicarbonate, Normal | 7
  Bicarbonate, High: number analyzed (Participants) | 11
  Bicarbonate, High | 2
  Lactate Dehydrogenase, Low: number analyzed (Participants) | 10
  Lactate Dehydrogenase, Low | 1
  Lactate Dehydrogenase, Normal: number analyzed (Participants) | 10
  Lactate Dehydrogenase, Normal | 7
  Lactate Dehydrogenase, High: number analyzed (Participants) | 10
  Lactate Dehydrogenase, High | 2
  Serum Total Protein, Low: number analyzed (Participants) | 11
  Serum Total Protein, Low | 3
  Serum Total Protein, Normal: number analyzed (Participants) | 11
  Serum Total Protein, Normal | 8
  Serum Total Protein, High: number analyzed (Participants) | 11
  Serum Total Protein, High | 0
  Low-Density Lipoprotein, Low: number analyzed (Participants) | 10
  Low-Density Lipoprotein, Low | 1
  Low-Density Lipoprotein, Normal: number analyzed (Participants) | 10
  Low-Density Lipoprotein, Normal | 2
  Low-Density Lipoprotein, High: number analyzed (Participants) | 10
  Low-Density Lipoprotein, High | 7
  High-Density Lipoprotein, Low: number analyzed (Participants) | 10
  High-Density Lipoprotein, Low | 6
  High-Density Lipoprotein, Normal: number analyzed (Participants) | 10
  High-Density Lipoprotein, Normal | 4
  High-Density Lipoprotein, High: number analyzed (Participants) | 10
  High-Density Lipoprotein, High | 0
  Thyroid-Stimulating Hormone, Low: number analyzed (Participants) | 9
  Thyroid-Stimulating Hormone, Low | 2
  Thyroid-Stimulating Hormone, Normal: number analyzed (Participants) | 9
  Thyroid-Stimulating Hormone, Normal | 6
  Thyroid-Stimulating Hormone, High: number analyzed (Participants) | 9
  Thyroid-Stimulating Hormone, High | 1
  T3, Low: number analyzed (Participants) | 9
  T3, Low | 2
  T3, Normal: number analyzed (Participants) | 9
  T3, Normal | 7
  T3, High: number analyzed (Participants) | 9
  T3, High | 0
  T4, Low: number analyzed (Participants) | 9
  T4, Low | 1
  T4, Normal: number analyzed (Participants) | 9
  T4, Normal | 7
  T4, High: number analyzed (Participants) | 9
  T4, High | 1

13. Secondary Outcome: Change From Baseline in QT Interval Corrected According to the Formula of Fridericia (QTcF), QT, QRS, and PR Duration
Description: Change from baseline in QTcF, QT, QRS, and PR duration were reported. QT interval is the time from electrocardiogram Q wave to the end of the T wave corresponding to electrical systole. QRS interval is the time from electrocardiogram Q wave to the end of the S wave, corresponding to ventricle depolarization. PR interval is the time between the beginning of the P wave and the start of the QRS interval, corresponding to the end of atrial depolarization and onset of ventricular depolarization.
Time Frame: Baseline, Day 15 of Cycle 1, 2, Day 1 of Cycle 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 (each cycle of 28 days), and End of treatment (up to 7 days after study treatment discontinuation)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
milliseconds
  QTcF: Baseline | 423.9 (24.84)
  QTcF: Change at Cycle 1, Day 15: number analyzed (Participants) | 7
  QTcF: Change at Cycle 1, Day 15 | 0.6 (16.11)
  QTcF: Change at Cycle 2, Day 1: number analyzed (Participants) | 7
  QTcF: Change at Cycle 2, Day 1 | 3.1 (28.33)
  QTcF: Change at Cycle 2, Day 15: number analyzed (Participants) | 4
  QTcF: Change at Cycle 2, Day 15 | -62.0 (99.90)
  QTcF: Change at Cycle 3, Day 1: number analyzed (Participants) | 5
  QTcF: Change at Cycle 3, Day 1 | 7.0 (14.30)
  QTcF: Change at Cycle 4, Day 1: number analyzed (Participants) | 3
  QTcF: Change at Cycle 4, Day 1 | 1.3 (11.50)
  QTcF: Change at Cycle 5, Day 1: number analyzed (Participants) | 3
  QTcF: Change at Cycle 5, Day 1 | 0.7 (1.53)
  QTcF: Change at Cycle 6, Day 1: number analyzed (Participants) | 3
  QTcF: Change at Cycle 6, Day 1 | -6.0 (9.17)
  QTcF: Change at Cycle 7, Day 1: number analyzed (Participants) | 2
  QTcF: Change at Cycle 7, Day 1 | -18.5 (6.36)
  QTcF: Change at Cycle 8, Day 1: number analyzed (Participants) | 1
  QTcF: Change at Cycle 8, Day 1 | -28.0 (NA) — Standard deviation was not estimated due to single participant.
  QTcF: Change at Cycle 9, Day 1: number analyzed (Participants) | 1
  QTcF: Change at Cycle 9, Day 1 | -36.0 (NA) — Standard deviation was not estimated due to single participant.
  QTcF: Change at Cycle 10, Day 1: number analyzed (Participants) | 1
  QTcF: Change at Cycle 10, Day 1 | -26.0 (NA) — Standard deviation was not estimated due to single participant.
  QTcF: Change at End of Treatment: number analyzed (Participants) | 8
  QTcF: Change at End of Treatment | 4.5 (25.69)
  QT: Baseline | 394.2 (36.19)
  QT: Change at Cycle 1, Day 15: number analyzed (Participants) | 7
  QT: Change at Cycle 1, Day 15 | -4.3 (18.27)
  QT: Change at Cycle 2, Day 1: number analyzed (Participants) | 7
  QT: Change at Cycle 2, Day 1 | -2.4 (29.47)
  QT: Change at Cycle 2, Day 15: number analyzed (Participants) | 5
  QT: Change at Cycle 2, Day 15 | -47.0 (79.97)
  QT: Change at Cycle 3, Day 1 | 6.6 (30.59)
  QT: Change at Cycle 4, Day 1: number analyzed (Participants) | 3
  QT: Change at Cycle 4, Day 1 | -6.7 (25.40)
  QT: Change at Cycle 5, Day 1: number analyzed (Participants) | 3
  QT: Change at Cycle 5, Day 1 | 5.3 (11.02)
  QT: Change at Cycle 6, Day 1: number analyzed (Participants) | 3
  QT: Change at Cycle 6, Day 1 | -6.7 (24.68)
  QT: Change at Cycle 7, Day 1: number analyzed (Participants) | 2
  QT: Change at Cycle 7, Day 1 | -33.0 (29.70)
  QT: Change at Cycle 8, Day 1: number analyzed (Participants) | 1
  QT: Change at Cycle 8, Day 1 | -78.0 (NA) — Standard deviation was not estimated due to single participant.
  QT: Change at Cycle 9, Day 1: number analyzed (Participants) | 1
  QT: Change at Cycle 9, Day 1 | -29.0 (NA) — Standard deviation was not estimated due to single participant.
  QT: Change at Cycle 10, Day 1: number analyzed (Participants) | 1
  QT: Change at Cycle 10, Day 1 | -18.0 (NA) — Standard deviation was not estimated due to single participant.
  QT: Change at End of Treatment: number analyzed (Participants) | 8
  QT: Change at End of Treatment | -0.3 (20.04)
  QRS: Baseline | 93.9 (12.75)
  QRS: Change at Cycle 1, Day 15: number analyzed (Participants) | 7
  QRS: Change at Cycle 1, Day 15 | -2.3 (4.68)
  QRS: Change at Cycle 2, Day 1: number analyzed (Participants) | 7
  QRS: Change at Cycle 2, Day 1 | -1.1 (13.50)
  QRS: Change at Cycle 2, Day 15: number analyzed (Participants) | 5
  QRS: Change at Cycle 2, Day 15 | 0.6 (6.31)
  QRS: Change at Cycle 3, Day 1: number analyzed (Participants) | 5
  QRS: Change at Cycle 3, Day 1 | -2.4 (2.61)
  QRS: Change at Cycle 4, Day 1: number analyzed (Participants) | 3
  QRS: Change at Cycle 4, Day 1 | -5.0 (3.61)
  QRS: Change at Cycle 5, Day 1: number analyzed (Participants) | 3
  QRS: Change at Cycle 5, Day 1 | -3.3 (3.06)
  QRS: Change at Cycle 6, Day 1: number analyzed (Participants) | 3
  QRS: Change at Cycle 6, Day 1 | 0.0 (4.00)
  QRS: Change at Cycle 7, Day 1: number analyzed (Participants) | 2
  QRS: Change at Cycle 7, Day 1 | -5.0 (1.41)
  QRS: Change at Cycle 8, Day 1: number analyzed (Participants) | 1
  QRS: Change at Cycle 8, Day 1 | -8.0 (NA) — Standard deviation was not estimated due to single participant.
  QRS: Change at Cycle 9, Day 1: number analyzed (Participants) | 1
  QRS: Change at Cycle 9, Day 1 | 5.0 (NA) — Standard deviation was not estimated due to single participant.
  QRS: Change at Cycle 10, Day 1: number analyzed (Participants) | 1
  QRS: Change at Cycle 10, Day 1 | 6.0 (NA) — Standard deviation was not estimated due to single participant.
  QRS: Change at End of Treatment: number analyzed (Participants) | 8
  QRS: Change at End of Treatment | -6.1 (6.01)
  PR: Baseline | 145.8 (25.13)
  PR: Change at Cycle 1, Day 15: number analyzed (Participants) | 7
  PR: Change at Cycle 1, Day 15 | -7.3 (19.60)
  PR: Change at Cycle 2, Day 1: number analyzed (Participants) | 7
  PR: Change at Cycle 2, Day 1 | -7.4 (26.50)
  PR: Change at Cycle 2, Day 15: number analyzed (Participants) | 5
  PR: Change at Cycle 2, Day 15 | 1.2 (11.37)
  PR: Change at Cycle 3, Day 1: number analyzed (Participants) | 5
  PR: Change at Cycle 3, Day 1 | -0.6 (19.59)
  PR: Change at Cycle 4, Day 1: number analyzed (Participants) | 3
  PR: Change at Cycle 4, Day 1 | -6.0 (2.00)
  PR: Change at Cycle 5, Day 1: number analyzed (Participants) | 3
  PR: Change at Cycle 5, Day 1 | 7.3 (16.29)
  PR: Change at Cycle 6, Day 1: number analyzed (Participants) | 3
  PR: Change at Cycle 6, Day 1 | 2.7 (21.39)
  PR: Change at Cycle 7, Day 1: number analyzed (Participants) | 2
  PR: Change at Cycle 7, Day 1 | 10.0 (22.63)
  PR: Change at Cycle 8, Day 1: number analyzed (Participants) | 1
  PR: Change at Cycle 8, Day 1 | -14.0 (NA) — Standard deviation was not estimated due to single participant.
  PR: Change at Cycle 9, Day 1: number analyzed (Participants) | 1
  PR: Change at Cycle 9, Day 1 | -13.0 (NA) — Standard deviation was not estimated due to single participant.
  PR: Change at Cycle 10, Day 1: number analyzed (Participants) | 1
  PR: Change at Cycle 10, Day 1 | -8.0 (NA) — Standard deviation was not estimated due to single participant.
  PR: Change at End of Treatment: number analyzed (Participants) | 8
  PR: Change at End of Treatment | -6.9 (21.96)

14. Secondary Outcome: Change From Baseline in Heart Rate
Description: Change from baseline in heart rate in terms of beats per minute was reported.
Time Frame: as for outcome 13
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | LGX818 (Encorafenib)
Number analyzed (Participants) | 12
beats per minute
  Baseline | 77.3 (15.79)
  Change at Cycle 1, Day 15: number analyzed (Participants) | 7
  Change at Cycle 1, Day 15 | 2.9 (9.01)
  Change at Cycle 2, Day 1: number analyzed (Participants) | 7
  Change at Cycle 2, Day 1 | 4.1 (12.31)
  Change at Cycle 2, Day 15: number analyzed (Participants) | 5
  Change at Cycle 2, Day 15 | -1.0 (9.30)
  Change at Cycle 3, Day 1: number analyzed (Participants) | 5
  Change at Cycle 3, Day 1 | -0.4 (12.66)
  Change at Cycle 4, Day 1: number analyzed (Participants) | 3
  Change at Cycle 4, Day 1 | 7.3 (14.74)
  Change at Cycle 5, Day 1: number analyzed (Participants) | 3
  Change at Cycle 5, Day 1 | -3.0 (5.29)
  Change at Cycle 6, Day 1: number analyzed (Participants) | 3
  Change at Cycle 6, Day 1 | -0.7 (7.77)
  Change at Cycle 7, Day 1: number analyzed (Participants) | 2
  Change at Cycle 7, Day 1 | 7.0 (11.31)
  Change at Cycle 8, Day 1: number analyzed (Participants) | 1
  Change at Cycle 8, Day 1 | 27.0 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 9, Day 1: number analyzed (Participants) | 1
  Change at Cycle 9, Day 1 | -2.0 (NA) — Standard deviation was not estimated due to single participant.
  Change at Cycle 10, Day 1: number analyzed (Participants) | 1
  Change at Cycle 10, Day 1 | -4.0 (NA) — Standard deviation was not estimated due to single participant.
  Change at End of Treatment: number analyzed (Participants) | 8
  Change at End of Treatment | 2.0 (10.68)

ADVERSE EVENTS:
Time Frame: From screening up to 30 days after the last dose of study treatment (maximum up to 13.3 months)
Description: Same event may appear as both AE and SAE. An event may be categorized as serious in 1 participant and non-serious in other, or participant may have experienced both SAE and non-SAE. The safety set included all participants who received at least one dose of study treatment and had at least one post-baseline safety assessment.
Arm/Group | LGX818 (Encorafenib)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LGX818 (Encorafenib) (N=12)
Anaemia (Blood and lymphatic system disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Fatigue (General disorders) | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LGX818 (Encorafenib) (N=12)
Anaemia (Blood and lymphatic system disorders) | 1
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Palpitations (Cardiac disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Conjunctival disorder (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Eye pruritus (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 4
Abdominal pain (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 3
Dyspepsia (Gastrointestinal disorders) | 1
Gastric fistula (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Retching (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 7
Asthenia (General disorders) | 3
Influenza like illness (General disorders) | 2
Mucosal inflammation (General disorders) | 2
Oedema peripheral (General disorders) | 2
Axillary pain (General disorders) | 1
Chills (General disorders) | 1
Face oedema (General disorders) | 1
Nodule (General disorders) | 1
Pyrexia (General disorders) | 1
Oral candidiasis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Candida infection (Infections and infestations) | 1
Folliculitis (Infections and infestations) | 1
Gastrointestinal infection (Infections and infestations) | 1
Electrocardiogram QT prolonged (Investigations) | 2
Weight decreased (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine decreased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Lipase increased (Investigations) | 1
Prothrombin time prolonged (Investigations) | 1
Urine leukocyte esterase (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Neoplasm skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 3
Headache (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 2
Dysaesthesia (Nervous system disorders) | 1
Narcolepsy (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Depression (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Glycosuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Micturition urgency (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Scrotal oedema (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Erythema (Skin and subcutaneous tissue disorders) | 3
Skin exfoliation (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 2
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Lentigo (Skin and subcutaneous tissue disorders) | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash follicular (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin burning sensation (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin tightness (Skin and subcutaneous tissue disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Due to slow enrollment and lack of response observed during the enrollment period, the Sponsor decided to close study enrollment early on 28 January 2015.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.